CLINICAL TRIAL: NCT03362372
Title: MEDISTAR STUDY: Mediterranean Diet and Smoking in Tarragona and Reus
Brief Title: Effect of the Mediterranean Diet on Lung Function in Smokers Without Previous Respiratory Disease
Acronym: MEDISTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SLT002/16/00155
Record Dates: First submitted 2017-10-09; First posted 2017-12-05 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Controlled, parallel, multicenter, cluster-randomized clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP: MEDITERRANEAN DIET COUNSELING (Experimental): During 2 years a nutritional intervention will be carried out to increase adherence to DiMet based on: annual visit of personalized nutritional education, a telephone contact for intervention reinforcement and computer access to a nutrition blog
  Interventions: Behavioral: Mediterranean diet counseling
- CONTROL GROUP: WITHOUT CHANGES IN DIET (No Intervention): The participants of health centers will carry out the same 5 visits (3 individual visits and 2 phone calls), although no changes are induced in their usual diet and they will not be offered access to the nutritional blog.

INTERVENTIONS:
Behavioral: Mediterranean diet counseling — The participants of the intervention CAP will enter into an educational program to increase adherence to the DiMet that will integrate three operational components:
  1. Explain the particularities of DiMet and the benefits of its monitoring. It will be an individual visit of 25-30 minutes (V1) where the study variables will be collected and the medical tests will be performed and repeated annually for two years (V3 and V5).
  2. Clarify the doubts of the DiMet monitoring and the advice received. It will be a telephone visit to reinforce the intervention, with annual frequency, for two years (V2 and V4).
  3. Report on DiMet's own foods, cooking habits, adapted recipes and other related topics. It will be for access to an ad hoc designed nutrition blog.
  Arms: INTERVENTION GROUP: MEDITERRANEAN DIET COUNSELING

SUMMARY:
Several studies have shown the influence of the eating pattern on lung function. However, the benefits of the Mediterranean diet (DiMet) in preventing pulmonary dysfunction are not well known.

Objective: To evaluate the effect of adherence to DiMet on the deterioration of lung function in smokers.

Methodology: Design: Controlled, parallel, multicenter, cluster-randomized clinical trial. Participants: 566 active smokers with a cumulative consumption of more than 10 packets a year, within 25 to 75 year-old age group, without previous respiratory disease and who agree with the conditions of the study and sign an informed consent . Scope: 20 Primary Care Centers managed by the Catalan Health Institutes in Tarragona that will be randomly assigned to a control or an intervention group (1: 1). Intervention: During 2 years a nutritional intervention will be carried out to increase adherence to DiMet based on: 1) annual visit of personalized nutritional education, 2) annual telephone contact for intervention reinforcement, and 3) computer access to a dietary block designed ad hoc. The control group will follow their usual diet style. All participants will receive advice to quit smoking. It will be evaluated: a) pulmonary function by forced spirometry and b) adherence to the DiMet with a questionnaire of 14 items and biological determinations. Statistical analysis: For intention to treat. The unit of analysis will be the individual smoker. Parameters of pulmonary function and adherence to the DiMet of both groups will be compared.

Expected results: DiMet prevents the appearance of altered lung function in smokers without previous respiratory pathology. Thus, DiMet will be key in pulmonary prevention, together with the fundamental recommendation of smoking cessation.

DETAILED DESCRIPTION:
Several studies have shown the influence of the eating pattern on lung function. However, the benefits of the Mediterranean diet (DiMet) in preventing pulmonary dysfunction are not well known.

Objective: To evaluate the effect of adherence to DiMet on the deterioration of lung function in smokers.

Methodology: Design: Controlled, parallel, multicenter, cluster-randomized clinical trial. Participants: 566 active smokers with a cumulative consumption of more than 10 packets a year, within 25 to 75 year-old age group, without previous respiratory disease and who agree with the conditions of the study and sign an informed consent . Scope: 20 Primary Care Centers managed by the Catalan Health Institutes in Tarragona that will be randomly assigned to a control or an intervention group (1: 1). Intervention: During 2 years a nutritional intervention will be carried out to increase adherence to DiMet based on: 1) annual visit of personalized nutritional education, 2) annual telephone contact for intervention reinforcement, and 3) computer access to a dietary block designed ad hoc. The control group will follow their usual diet style. All participants will receive advice to quit smoking. It will be evaluated: a) pulmonary function by forced spirometry and b) adherence to the DiMet with a questionnaire of 14 items and biological determinations. Statistical analysis: For intention to treat. The unit of analysis will be the individual smoker. Parameters of pulmonary function and adherence to the DiMet of both groups will be compared.

Expected results: DiMet prevents the appearance of altered lung function in smokers without previous respiratory pathology. Thus, DiMet will be key in pulmonary prevention, together with the fundamental recommendation of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Active smoking and cumulative consumption ≥10 pack-years.
* Age between 25-75 years.
* Internet connection.

Exclusion Criteria:

* History of respiratory disease.
* Chronic or terminal disorder that alters basal parameters.
* Any reason that limits follow up.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in lung function values in smokers without previous respiratory disease | 2 years
  Changes in lung function measured by spirometry. An altered lung function was considered if values of FVC <80% and / or FEV1 <80% and / or FEV1 / FVC <0.7

SECONDARY OUTCOMES:
Nutritional intervention | 2 years
  The effectiveness of the intervention will be measured by dietary changes by a food frequency questionnaire
Nutritional intervention | 2 years
  Adherence to the Mediterranean diet will be measured by dietary changes in a mediterranean diet adherence score of 14-ítem
Anthropometric parameters | 2 years
  Changes in anthropometric parameters: weight in kilograms and height in meters. Weight and height will be combined to report BMI in kg/m2
Anthropometric parameters | 2 years
  Changes in anthropometric parameters: abdominal perimeter
Changes in food consumption markers | 2 years
  Changes in food consumption markers: excreted of total polyphenols in fresh urine.
Changes in inflammation markers | 2 years
  Changes in serum inflammation markers: high-sensitivity C-reactive protein
Changes in inflammation markers | 2 years
  Changes in serum inflammation markers: interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Martín Luján, Principal Investigator — Catalan Institute of Health
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Spain

REFERENCES:
- [Result] Martin-Lujan F, Catalin RE, Salamanca-Gonzalez P, Sorli-Aguilar M, Santigosa-Ayala A, Valls-Zamora RM, Martin-Vergara N, Canela-Armengol T, Arija-Val V, Sola-Alberich R. A clinical trial to evaluate the effect of the Mediterranean diet on smokers lung function. NPJ Prim Care Respir Med. 2019 Nov 27;29(1):40. doi: 10.1038/s41533-019-0153-7. PMID 31776344
- [Result] Catalin RE, Martin-Lujan F, Salamanca-Gonzalez P, Palleja-Millan M, Villalobos F, Santigosa-Ayala A, Pedret A, Valls-Zamora RM, Sola R, On Behalf Of The Medistar Research Group Investigators. Mediterranean Diet and Lung Function in Adults Current Smokers: A Cross-Sectional Analysis in the MEDISTAR Project. Nutrients. 2023 Mar 3;15(5):1272. doi: 10.3390/nu15051272. PMID 36904270

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03362372/Prot_SAP_ICF_000.pdf